CLINICAL TRIAL: NCT00724477
Title: PRAGMATIC (This is the True Official Title of the Protocol for This Study)
Brief Title: Retrospective Evaluation of the Percentage of Subjects Who Have Reached Their LDL-C Objectives After Treatment With INEGY (Study P05103)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05103
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects treated with INEGY: Subjects suffering from primary hypercholesterolemia that are not controlled by statins as a monotherapy, and are treated with INEGY
  Interventions: Drug: INEGY

INTERVENTIONS:
Drug: INEGY — Ezetimibe 10mg - Simvastatine 20 mg or 40 mg; Tablet - OD; Patient currently treated for INEGY for at least 4 weeks
  Other Names: SCH 465981

SUMMARY:
The main objective of this study is to determine the percentage of patients who met the low-density lipoprotein cholesterol (LDL-C) objective with INEGY, that were not under statin monotherapy treatment.

DETAILED DESCRIPTION:
The type of patient sampling used was consecutive patient sampling

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged over 18;
* patient suffering from primary hypercholesterolemia;
* patient justifying treatment with INEGY® (2nd intention);
* patient currently treated with INEGY® for at least 4 weeks;
* patient with a lipid profile before treatment with INEGY®, documenting a level of LDL-C exceeding the therapeutic objective under treatment with a statin as monotherapy;
* patient with an evaluation of lipid disorder (EAL) treated with INEGY®, performed within 1 to 3 months of starting treatment.

Exclusion Criteria:

* patient not previously treated with a statin;
* patient previously treated with a combination of hypolipemics;
* patient treated with INEGY® as first intention;
* patient treated with INEGY® for less than 4 weeks;
* patient already included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from primary hypercholesterolemia that are not controlled by statins as a monotherapy, and are treated with INEGY
Sampling Method: Probability Sample
Enrollment: 1663 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Treated With INEGY: Subjects suffering from primary hypercholesterolemia that were not adequately controlled by statins as a monotherapy, and were treated with INEGY. INEGY is composed of a combination of ezetimibe (10 mg) and simvastatin (20 or 40 mg). The dosage of the study treatment is one tablet per day ezetimibe/simvastatin (10 mg/20 mg or 10 mg/40 mg).
Period: Overall Study
Arm/Group | Subjects Treated With INEGY
Started | 1663 (This safety population (SAF)analysed consisted of all patients who took at least one tablet of INEGY)
Completed | 1663
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Treated With INEGY
Number analyzed (Participants) | 1663
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 585
  Male | 1078
Region of Enrollment [Number; unit: participants]
  France | 1663

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching the Targeted LDL-C Levels
Description: A subject was considered to have met targeted LDL-C levels (been controlled) if:
  * subject had no cardiovascular (CV) risk factors and level of LDL-C after initiating INEGY was lower than 2.2 g/L,
  * subject had only 1 CV risk factor and level of LDL-C after initiating INEGY was lower than 1.9 g/L,
  * subject had 2 CV risk factors and level of LDL-C after initiating INEGY was lower than 1.6 g/L,
  * subject had 3 or more CV risk factors and level of LDL-C after initiating INEGY was lower than 1.3 g/L,
  * subject had a high CV risk and level of LDL-C after initiating INEGY was lower than 1 g/L.
Time Frame: 1 to 3 months after starting treatment
Population: This was the efficacy population per protocol (PP) targeted for study treatment, and consisted of patients having taken INEGY at least once, with a primary efficacy criterion available (presence of risk factors or not plus lipid assessment after introduction of INEGY), and showing no major deviations from the protocol.
Measure: Number; unit: Participants
Arm/Group | Subjects Treated With INEGY
Number analyzed (Participants) | 1354
Participants | 740

ADVERSE EVENTS:
Time Frame: 4 weeks to 3 months
Description: Adverse events were recorded from the introduction of INEGY to the first assessment after introduction of INEGY
Arm/Group | Subjects Treated With INEGY
Serious Adverse Events (participants affected / at risk) | 2/1663
Other Adverse Events (participants affected / at risk) | 0/1663
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Treated With INEGY (N=1663)
Myocardial infarction (Endocrine disorders) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this non-interventional study can be published or presented by members of the scientific committee after revision and agreement by Schering-Plough, and in such a way that the confidential information and industrial property are not revealed. Before publication or presentation, a copy of the final text must be sent by the member(s) of the scientific committee to Schering-Plough for comment.